CLINICAL TRIAL: NCT01156545
Title: A Randomized Open Label Phase II Trial Comparing BIBW2992 Plus Simvastatin With BIBW2992 Plus Best Supportive Care in Previously Treated Patients With Advanced (Stage IIIB/IV) Non-adenocarcinomatous Non-small Cell Lung Cancer (NSCLC)
Brief Title: BIBW 2992 Plus Simvastatin vs. BIBW 2992 in Previously Treated Patients With Advanced Non-adenocarcinomatous NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-489; BIBW 2992 1200.113 (Other: Boehringer-ingelheim protocol number)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: BIBW 2992; Simvastatin; NSCLC; advanced stage; previously treated patients; non-adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm (Experimental): BIBW 2992 plus simvastatin arm
  Interventions: Drug: BIBW 2992; Drug: simvastatin
- control arm (Active Comparator): BIBW 2992 arm
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — BIBW 2992 40mg, once a day, oral intake, every day
  Other Names: afatinib
Drug: simvastatin — simvastatin 40mg, once a day, oral intake, every day.
  Other Names: simvastar
  Arms: Treatment arm

SUMMARY:
The investigators hypothesized that simvastatin may enhance sensitivity to BIBW 2992 in non-adenocarcinoma that is relatively resistant to TKIs. Based on these data, the investigators will research the effectiveness comparing BIBW2992, an irreversible EGFR-TKI, plus simvastatin with BIBW2992 alone in the setting of a randomized phase II study in previously treated patients with advanced non-adenocarcinomatous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
One of the main reasons of resistance to EGFR tyrosine kinase inhibitors (TKIs) is that there are alternative mechanisms for persistent activating EGFR downstream signaling, including both RAS/Erk and PI3K/Akt kinase pathways. Therefore, simultaneous inhibition of both pathways would be necessary to reduce tumor cell survival more effectively. One of the candidate combinations is concurrent use of EGFR-TKIs and statins, which are irreversible inhibitors of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase and have been used to treat hypercholesterolemia through blocking the mevalonate biosynthesis pathway. Beside the cholesterol lowering effect, statins have been shown to induce apoptosis in several tumor types. It affects the synthesis of other products of the mevalonate pathway such as isoprenoids, which are used as substrates for prenylation. Attachment of isoprenoids to RAS proteins facilitates their anchoring to the cell membrane where they carried out their roles. By interrupting the biosynthesis of mevalonate, statins inhibit activation of RAS and downstream signaling cascades, including the RAF/MEK/ERK and PI3K/AKT, which play critical roles in regulation of cell survival and proliferation. Therefore, it seems to be a promising therapeutic approach overcoming tumor resistance to EGFR-TKIs, which is associated with RAS activation.

According to the recent clinical result of phase II trial, a randomized phase II study of gefitinib with or without simvastatin in previously treated patients with advanced NSCLC conducted by Han et al.37 gefitinib plus simvastatin combination produced higher response rates than gefitinib alone in patients with non-adenocarcinoma (5/13 [39%] v 1/13 [8%], P=0.06). This finding suggests that simvastatin may enhance sensitivity to gefitinib in non-adenocarcinoma that is relatively resistant to gefitinib. Moreover, by Mantha et al.35 demonstrated that the combination of gefitinib and lovastatin showed significant synergic cytotoxic effects in vitro in a total of 16 squamous cell carcinomas, NSCLC, and colon carcinoma cell lines. Of special interest, these cell lines did not possess the activating mutations of EGFR, which confer increased sensitivity to gefitinib. Nevertheless, combining lovastatin with gefitinib induced more significant inhibition of AKT activation than either agent alone. Additionally, lovastatin significantly enhanced the sensitivity to gefitinib treatment regardless PTEN loss in glioblastoma cell lines. These results suggest that statins can augment EGFR inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of Stage IIIB or Stage IV non-adenocarcinomatous non-small cell lung cancer (e.g., squamous cell or large cell carcinoma).(The 7th edition of the TNM classification for lung cancer47-See Appendix 6)
2. Progressive disease following the first or second line cytotoxic chemotherapy regimen(s) including at least one platinum-containing regimen.
3. Measurable disease according to RECIST 1.1.40
4. Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2.41
5. Age ≥ 18 years.
6. Life expectancy of at least three (3) months.
7. Written informed consent that is consistent with ICH-GCP guidelines.

Exclusion Criteria:

1. More than three (3) prior cytotoxic chemotherapy treatment regimen for relapsed or metastatic NSCLC.
2. Prior treatment with EGFR targeting small molecules or antibodies (e.g., gefitinib, erlotinib, cetuximab).
3. Chemotherapy, hormonal therapy (other than megestrol acetate or steroids required for maintenance non-cancer therapy), immunotherapy or surgery (other than biopsy) within 4 weeks prior to study entry.
4. Radiotherapy within 2 weeks prior to study entry. Only palliative radiotherapy to non-target lesion should be allowed for the entered cases.
5. Active brain metastases with clinically significant neurological symptoms or signs. Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs.
6. Any other current malignancy or malignancy diagnosed within the past five (5) years (other than non-melanomatous skin cancer and in situ cervical cancer).
7. Known pre-existing interstitial lung disease.
8. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g. Crohn's disease, malabsorption or CTC grade ≥2 diarrhea of any etiology.
9. Absolute neutrophil count (ANC) <1500 / mm3.
10. Platelet count < 100,000 / mm3.
11. Serum creatinine >1.5 times upper limit of normal (ULN) or creatinine clearance < 60 ml / min
12. Bilirubin > 1.5 times upper limit of normal.
13. Aspartate amino transferase (AST) or alanine amino transferase (ALT) > 3 times the upper limit of normal (ULN) (if related to liver metastases > 5 times ULN).
14. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to study entrance.
15. Cardiac left ventricular function with resting ejection fraction of less than 50%.
16. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
17. Women of childbearing potential, or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial.
18. Pregnancy or breast-feeding.
19. Patients unable to comply with the protocol.
20. Active hepatitis B infection, active hepatitis C infection or known HIV carrier.
21. Known or suspected active drug or alcohol abuse.
22. Requirement for treatment with any of the prohibited concomitant medications listed in Section 4.2.2.
23. Any contraindications for therapy with simvastatin.
24. Known hypersensitivity to BIBW 2992 or the excipients of any of the trial drugs.
25. Use of any investigational drug within 4 weeks of randomization (unless a longer time period is required by local regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate | each 8 weeks
  Repeat tumor assessments will be performed after the completion of Week 4, Week 8, and in 8-week intervals thereafter until progression or withdrawal for another reason

SECONDARY OUTCOMES:
Disease Control Rate | every 8 weeks
  Repeat tumor assessments will be performed after the completion of Week 4, Week 8, and in 8-week intervals thereafter until progression or withdrawal for another reason
Progression-Free Survival | every 8 weeks
  Repeat tumor assessments will be performed after the completion of Week 4, Week 8, and in 8-week intervals thereafter until progression or withdrawal for another reason
Overall Survival | every 12 weeks
  Overall survival (OS) will be calculated as the duration from the date of randomization to the date of disease progression or death, whichever occurs first.
Adverse event | first drug intake until 28 days after last treatment administration
  For grading of adverse events CTC AE criteria (version 4.0) will be utilizedStatistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events. To this end, all adverse events occurring between first drug intake until 28 days (inclusive) after last treatment administration will be considered 'treatment-emergent'. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.
Pharmacogenetic and biomarkers analyses | every 8 weeks
  The primary focus of predictive biomarker analyses is to investigate potential relationships of certain biomarkers with efficacy or safety endpoints. For this study, predictive efficacy analyses will be performed with such biomarkers as EGFR mutation status. EGFR mutation status will be measured in tumor samples and blood samples. In addition, plasma levels of IGFBP-3 and amphiregulin as well as gene polymorphisms related to the EGFR and IGF-1R pathways will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: JI-YOUN HAN, M.D. PhD., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea